CLINICAL TRIAL: NCT00171509
Title: A Multicenter, Randomized Open-label Pilot Study to Explore the Benefit of a Conversion From a Twice a Day Administration of Cyclosporine Microemulsion to a Once a Day Administration and to Identify the C2 Ranges to Target After Conversion in Stable Liver Transplant Recipients
Brief Title: Efficacy and Safety of Cyclosporine Microemulsion Given Once a Day in Adult Stable Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: COLO400A2421
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Liver Transplant
Keywords: Liver transplant, adults, once a day administration, Immunosuppressants

ARMS (3):
- BID cyclosporine (Active Comparator): control group continuing with a BID administration of cyclosporine and C2 monitoring.
  Interventions: Drug: Cyclosporine microemulsion
- OAD cyclosporine (Experimental): conversion to OAD administration of cyclosporine with the same daily dose as received prior to conversion
  Interventions: Drug: Cyclosporine microemulsion
- OAD cyclosporine reduced (Experimental): OAD administration of cyclosporine with a daily dose adjusted to a reduced C2
  Interventions: Drug: Cyclosporine microemulsion

INTERVENTIONS:
Drug: Cyclosporine microemulsion

SUMMARY:
The purpose of this study is to determine whether cyclosporine microemulsion given once a day instead of twice a day benefits kidney function, blood pressure, lipid profile and glucose control in stable liver transplant recipients. The study also aims to identify the target ranges of levels of cyclosporine microemulsion in the blood.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months post-transplant
* At least one of the following: stable or deteriorating kidney function, high blood pressure, high lipids, high glucose
* Receiving stable doses of cyclosporine microemulsion for the past 3 months

Exclusion Criteria:

* - Severe rejection within the past 3 months
* Severe kidney dysfunction
* Transplanted for hepatitis C or autoimmune hepatitis

Other protocol-defined exclusion criteria applied

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Investigation of the proportion of patients with an improving GFR in the groups converted to OAD in comparison with the BID group 15 weeks after conversion.

SECONDARY OUTCOMES:
assess the safety of a once a day administration of cyclosporine microemulsion.
compare for each patient the C2 levels pre- and post-conversion.
characterize the steady state pharmacokinetics of cyclosporine after conversion to once a day administration.
the proportion of patients with improving renal function or blood pressure or lipid levels or glucose control (as a composite end point as well as each parameter assessed individually) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis